CLINICAL TRIAL: NCT05831306
Title: A Randomized Clinical Trial Evaluating Two Different Diets for IBS
Brief Title: A Clinical Trial Evaluating Diets for IBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020P000625
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: dietary intervention; lifestyle intervention
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet A (Experimental): Modified Diet A
  Interventions: Other: Diet A
- Diet B (Experimental): Modified Diet B
  Interventions: Other: Diet B

INTERVENTIONS:
Other: Diet A — Modified Diet A
  Arms: Diet A
Other: Diet B — Modified Diet B
  Arms: Diet B

SUMMARY:
Diet and lifestyle changes are the recommended first line treatments for symptom relief in irritable bowel syndrome (IBS). Currently the only diet that is widely recommended and for which there is good evidence of efficacy in IBS is one low in fermentable oligosaccharides, disaccharides, monosaccharides, and polyols (low-FODMAP). While effective, the Low-FODMAP diet is burdensome and costly to patients and in clinical practice adherence to FODMAP restriction is less than optimal. Further, patients who respond to a FODMAP restriction often are reluctant to reintroduce more FODMAPs into their diet, which may deprive them of foods, particularly fruits and vegetables with important health benefits. Therefore, there is a need for other dietary interventions for IBS that are less burdensome to patients. This clinical trial assesses the efficacy of two dietary interventions.

ELIGIBILITY:
Inclusion criteria

1. Patients with IBS-D diagnosed per Rome IV questionnaire and without any unexplained alarm features (rectal bleeding, weight loss, nocturnal symptoms, family history of inflammatory bowel disease or celiac disease)
2. Aged 18-65 years at the time of screening
3. Weekly average of worst daily (in the past 24 hours) abdominal pain score of ≥3.0 on a 0- to-10 point scale
4. At least 80% compliance in daily diary entries during the 7-day screening period

Exclusion criteria

1. Subjects adhering to a dietary IBS-treatments such as the low-fat diet, low FODMAP diet, or gluten-free diet within the past 6 months
2. Subjects with a known food allergy to eggs, peanuts, or milk (subjects with lactose intolerance who are experiencing IBS symptoms while on a lactose-free diet will not be excluded from the study).
3. Subjects with a history of insulin-dependent or non-insulin-dependent diabetes
4. Subjects with a known history of celiac disease, inflammatory bowel disease or microscopic colitis
5. Subjects with a history of an eating disorder requiring medical or behavioral treatment within the past 10 years.
6. BMI < 18.5

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Abdominal Pain Intensity | 28 days
  Proportion of weekly responders. A weekly responder is defined as a decrease in weekly average of worst abdominal pain in the past 24 hours score of at least 30% compared with baseline.

SECONDARY OUTCOMES:
Abdominal Discomfort Intensity | 28 days
  Proportion of weekly responders. A weekly responder is defined as a decrease in worst abdominal discomfort in the past 24 hours score of at least 30% compared with baseline.
Composite Score | 28 days
  Proportion of weekly composite responders. A weekly composite responder is defined as a subject who experiences a decrease in the weekly average of worst abdominal pain in the 24 hours score of at least 30% compared with baseline AND who experiences a 50% or greater reduction in the number of days per week with at least one stool that has a consistency of Type 6 or 7 compared with baseline
Abdominal Bloating Intensity | 28 days
  Proportion of weekly responders. A weekly responder is defined as a decrease in worst abdominal bloating in the past 24 hours score of at least 30% compared with baseline.
Stool Consistency | 28 days
  Weekly responder. A weekly responder is defined as a decrease of at least 50% in the number of days per week with at least one stool that has a consistency of Bristol Stool Form Scale Type 6 or Type 7 compared with baseline.
Irritable Bowel Syndrome - Symptom Severity Score | 28 days
  Proportion of subjects who experience a 50-point and 100-point decrease in IBS-SSS compared with baseline.
Irritable Bowel Syndrome - Symptom Severity Score | 28 days
  Change in IBS-SSS as compared with baseline.
Adequate Relief | 28 days
  Proportion of subjects who experience adequate relief compared with baseline.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan - Ann Arbor, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh P, Chey SW, Nee J, Eswaran S; Dietary Therapy in IBS Working Group; Lembo A, Chey WD. Is a Simplified, Less Restrictive Low FODMAP Diet Possible? Results From a Double-Blind, Pilot Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2025 Feb;23(2):362-364.e2. doi: 10.1016/j.cgh.2024.04.021. Epub 2024 May 9. PMID 38729393